CLINICAL TRIAL: NCT05136469
Title: Comparison of Sciatic Nerve Gliding and Lower Extremity Dynamic Stretch on Hamstring Flexibility of Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/0401 Nasrullah
Record Dates: First submitted 2021-09-27; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEURAL GLIDING (Experimental): with Sciatic nerve gliding which is done by applying force on the proximal point and releasing the force distally and then reversing the process. This process was achieved for 30 seconds, 6 times on each leg for a total time of 3 minutes (360 seconds).
  Interventions: Other: NEURAL GLIDING
- DYNAMIC STRETCH (Active Comparator): The stretch force was applied on the ankle in downward direction which was held for 30 seconds and was repeated 5 times total of 2.5 minutes (150 seconds). Stretch was given on both legs one at a time. Treatment was given for 3 weeks with 2 sessions per week
  Interventions: Other: DYNAMIC STRETCH

INTERVENTIONS:
Other: NEURAL GLIDING — with Sciatic nerve gliding which is done by applying force on the proximal point and releasing the force distally and then reversing the process. This process was achieved for 30 seconds, 6 times on each leg for a total time of 3 minutes (360 seconds).
  Arms: NEURAL GLIDING
Other: DYNAMIC STRETCH — The stretch force was applied on the ankle in downward direction which was held for 30 seconds and was repeated 5 times total of 2.5 minutes (150 seconds). Stretch was given on both legs one at a time. Treatment was given for 3 weeks with 2 sessions per week
  Arms: DYNAMIC STRETCH

SUMMARY:
In this research, the main purpose is to determine the comparison of acute effect of sciatic nerve gliding and lower extremity dynamic stretching exercises on hamstring flexibility and athletic performance. The participants will be begin with warm-up sessions for 3-5 minutes then baseline data (pre-test): hamstring flexibility will be measured. The order of pre-test will be randomized and same order will be used for post-test. This is a community service addition, added so that everyone in the society can get to know the effects of nerve gliding and lower extremity dynamic stretches on hamstring flexibility, will be cost effective, and will reduce their visits to the therapist.

Randomized controlled trial with 1 month follow-up. The sample size is 40. subjects will be divided in two groups, 20 athletes will be given a session of sciatic nerve gliding while lower extremity stretch will be given to remaining 20 athletes. Study duration is of 6 months.Sampling technique employed will be convenient with random assignment. Individuals of age group 18-40 years having male gender regularly exercise at least once a week for 30 minutes. Tools used in the study are Universal inclinometer and Active knee extension test and SLR TEST. Data will be analyzed through IBM SPSS 23

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 year
* Footballers players
* Male gender
* Hamstring tightness of one or both legs,
* Unable to achieve greater than 160 degree of knee extension with hip at 90 degree of flexion
* Able to reach <70 degree hip flexion in SLR

Exclusion Criteria:

* Individuals who had sustained injury in the prior six months to the lumbar region,
* Limited activity level for more than 3 days,
* Low back problems (disc bulge etc.)
* Individual with a history of fracture or trauma were excluded from the study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Range of Hamstrings (Universal Goniometer) | 3 WEEKS
  Participants were asked to do SLR and active knee extensions and then measure range of hamstrings and then note the range by goniometer .
SLR test | 3 WEEKS
  Participants were asked to lie down in a supine position and were asked to raise their both leg one by one. In order to measure hamstring flexibility center of the goniometer was placed at the greater trochanter level its proximal arm at midline of pelvis and distal arm along the shaft of the femur referring lateral epicondyle. After which scoring were noted in which >110 showed excellent scoring, 80 to 110 showed good scoring and 60 to 79 showed fair scoring of the hamstring muscle flexibility
Knee Extension test | 3 WEEKS
  For active knee extension test participant one leg is vertically extended and the other leg was flexed on the level of hip joint and then the participants was asked to extend the knee. The point where the vertical leg starts to move is recorded. The angle between the thighs is measured, if the knee was fully extended it was noted as 0 and if it shows slight flexion that was noted as positive number like 20 or 30 degree. By following the same protocol both right and left legs were recorded. Normal knee extension ranges from 130_140 to 0 degree knee extension less than the range was written as negative number

CONTACTS AND LOCATIONS:
Overall Officials: sidra shafique, tDPT, Study Chair — RIU lahore
Locations (1):
- Pcb Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baxter C, Mc Naughton LR, Sparks A, Norton L, Bentley D. Impact of stretching on the performance and injury risk of long-distance runners. Res Sports Med. 2017 Jan-Mar;25(1):78-90. doi: 10.1080/15438627.2016.1258640. Epub 2016 Dec 2. PMID 27912252
- [Background] Castellote-Caballero Y, Valenza MC, Martin-Martin L, Cabrera-Martos I, Puentedura EJ, Fernandez-de-Las-Penas C. Effects of a neurodynamic sliding technique on hamstring flexibility in healthy male soccer players. A pilot study. Phys Ther Sport. 2013 Aug;14(3):156-62. doi: 10.1016/j.ptsp.2012.07.004. Epub 2012 Nov 8. PMID 23142014
- [Background] Lumbroso D, Ziv E, Vered E, Kalichman L. The effect of kinesio tape application on hamstring and gastrocnemius muscles in healthy young adults. J Bodyw Mov Ther. 2014 Jan;18(1):130-8. doi: 10.1016/j.jbmt.2013.09.011. Epub 2013 Oct 2. PMID 24411161
- [Background] Bonser RJ, Hancock CL, Hansberger BL, Loutsch RA, Stanford EK, Zeigel AK, Baker RT, May J, Nasypany A, Cheatham S. Changes in Hamstring Range of Motion After Neurodynamic Sciatic Sliders: A Critically Appraised Topic. J Sport Rehabil. 2017 Jul;26(4):311-315. doi: 10.1123/jsr.2015-0166. Epub 2016 Aug 24. PMID 27632844
- [Background] Kulendran T, Rajesh D, Kumar S. The Effect of One-Time Dynamic Soft Tissue Mobilization on Hamstring Flexibility Sustenance between Healthy Males and Females. Indian Journal of Public Health Research & Development. 2018;9(10).
- [Background] Fransson P, Johansson R, Hafstrom A, Magnusson M. Methods for evaluation of postural control adaptation. Gait Posture. 2000 Sep;12(1):14-24. doi: 10.1016/s0966-6362(00)00052-7. PMID 10996293